CLINICAL TRIAL: NCT05064345
Title: A Phase Ia, Randomized, Double-blind, Placebo-controlled, Single Dose-escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HB0034 in Adult Healthy Subjects
Brief Title: A Study to Evaluate HB0034 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HB0034-01
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- HB0034 dose group 1 (Active Comparator): HB0034 single dose
  Interventions: Drug: HB0034
- HB0034 dose group 2 (Active Comparator): HB0034 single dose
  Interventions: Drug: HB0034
- HB0034 dose group 3 (Active Comparator): HB0034 single dose
  Interventions: Drug: HB0034
- HB0034 dose group 4 (Active Comparator): HB0034 single dose
  Interventions: Drug: HB0034
- HB0034 dose group 5 (Active Comparator): HB0034 single dose
  Interventions: Drug: HB0034
- HB0034 dose group 6 (Active Comparator): HB0034 single dose
  Interventions: Drug: HB0034
- HB0034 dose group 7 (Active Comparator): HB0034 single dose
  Interventions: Drug: HB0034
- Matching placebo for each dose group (Placebo Comparator): placebo, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HB0034 — Recombinant Humanized Anti-IL-36R Monoclonal antibody
  Other Names: no other invention names
  Arms: HB0034 dose group 1; HB0034 dose group 2; HB0034 dose group 3; HB0034 dose group 4; HB0034 dose group 5; HB0034 dose group 6; HB0034 dose group 7
Drug: Placebo — Palcebo
  Other Names: no other invention names
  Arms: Matching placebo for each dose group

SUMMARY:
The aim of this study is to investigate the safety and tolerability of HB0034 in healthy subjects following a single dose.

DETAILED DESCRIPTION:
This is a first-in-human (FIH) study of HB0034 to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of HB0034.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects age ≥ 18 and ≤ 55 years.
* Body Mass Index (BMI) ≥ 17.5 and ≤ 32 kg/m².
* Normal ECG, blood pressure, respiratory rate, temperature, and heart rate, unless the investigator considers any abnormality to be not clinically significant.
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation.

Exclusion Criteria:

* History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease.
* Current or history of malignancy.
* Family history of premature Coronary Heart Disease (CHD)
* History of clinically significant opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia).
* Pregnant or Breasting feeding subject. Women with a positive pregnancy test (HCG).
* Further exclusions criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with drug related adverse events (AEs) | up to 2000 hours
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational drug

SECONDARY OUTCOMES:
Cmax | up to 2000 hours
  The maximum measured concentration of the analysis in plasma

OTHER OUTCOMES:
AUC0-infinity | up to 2000 hours
  The area under the concentration-time curve of the analysis in plasma over the time interval from 0 extrapolated to infinity

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schwabe, Principal Investigator — NZCR OpCo limited AKL
Locations (1):
- New zealand Clinical Research, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No